CLINICAL TRIAL: NCT00512187
Title: Moderate Weight Loss Makes Obese Patients With Severe Chronic Plaque Psoriasis Responsive to Sub-Optimal Dose of Cyclosporine: an Investigator Blinded, Controlled, Randomized Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita di Verona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GISONDI 1; no grants received at all
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2007-08-07 (Estimated); Status verified 2007-08

CONDITIONS: Chronic Plaque Psoriasis; Obesity
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- first group (Experimental): patients who adhered to a low-calorie diet associated to sub-optimal cyclosporine dose (2.5 mg/Kg/day)for 24 weeks
  Interventions: Other: low calorie diet

INTERVENTIONS:
Other: low calorie diet — Low calorie diet was designed to achieve a loss of 5-10% of initial weight. All enrolled patients received a balanced diet scheme, based on a caloric intake reduction related to BMI and sex (range 1200-1500 Kcal/day for women, 1300-1600 Kcal/day for men). Calorie intake consisted approximately of 60% carbohydrates, 25% fat, 15% protein

SUMMARY:
The study hypothesis is to investigate whether a moderate weight loss (i.e. a weight reduction of at least 5%) could improve the response rate to a suboptimal dose of cyclosporine in patients with severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age,active but clinically stable plaque psoriasis involving at least 10 percent of the body surface area and a psoriasis area and severity index (PASI) score ≥10 and a body mass index ≥30.

Exclusion Criteria:

* Other type of psoriasis (guttate, erythrodermic and pustular psoriasis)
* Uncontrolled hypertension
* Severe congestive heart failure
* Renal and liver impairment
* Active or chronic infections, including HIV, HBV and HCV infections, latent tuberculosis
* Previous or active malignancies
* Pregnancy and lactations
* Previous treatment with cyclosporine
* Phototherapy or any systemic or topical therapy for psoriasis within the previous 4 weeks before enrolment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-11; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Primary end point PASI 75 response | week 24

SECONDARY OUTCOMES:
secondary end point was % of body weight reduction | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Giampiero Girolomoni, Principal Investigator — University of Verona, Section of Dermatology and Venereology
Locations (1):
- University of Verona, Verona, Italy

REFERENCES:
- [Derived] Gisondi P, Del Giglio M, Di Francesco V, Zamboni M, Girolomoni G. Weight loss improves the response of obese patients with moderate-to-severe chronic plaque psoriasis to low-dose cyclosporine therapy: a randomized, controlled, investigator-blinded clinical trial. Am J Clin Nutr. 2008 Nov;88(5):1242-7. doi: 10.3945/ajcn.2008.26427. PMID 18996858